CLINICAL TRIAL: NCT06503445
Title: The Impact of Video-based Cardiac Rehabilitation Education in Patients With Cardiovascular Implantable Electronic Devices(CIEDs)- a Randomized Controlled Trial
Brief Title: The Impact of Video-based Cardiac Rehabilitation Education in Patients With CIEDs- a Randomized Controlled Trial
Acronym: CIEDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109-064-E
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Patients With Cardiac Implantable Electronic Devices
Keywords: Cardiac implantable electronic device; cardiac rehabilitation; video-based education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The experimental group with cardiac implantable electronic devices will receive cardiac rehabilitation health education video intervention.
  Interventions: Other: education video
- Control group (Sham Comparator): The control group with cardiac implantable electronic devices will receive only health education video intervention.
  Interventions: Other: education video

INTERVENTIONS:
Other: education video — the intervention group will watch the cardiac reahbiltation health education video.
  the control group will watch the health educatopm video.

SUMMARY:
Cardiac rehabilitation has the beneficial effects of secondary prevention and social psychological and physical health status in patients with cardiovascular diseases. International and clinical guidelines currently recommend exercise training and rehabilitation for heart failure patients, which can effectively improve mortality and prognosis. However, few of these recommendations have specific recommendations for patients with cardiac implantable electronic devices. Currently the recommendations of cardiac rehabilitation include patients with coronary heart disease (acute coronary heart disease, any coronary revascularization, stable coronary disease or unstable angina), patients with heart failure, after cardiac surgery, and patients with high cardiovascular risk. Many of these patients may be implanted with cardiac implantable electronic devices. In 2011, 938 pacemakers, 140 cardiac resynchronization therapy and 149 implantable cardioverter defibrillators were implanted per million inhabitants in Europe. Therefore, among the groups with cardiac implantable electronic devices, cardiac rehabilitation plays a certain role. The purpose of this study is to evaluate whether video-based cardiac rehabilitation health education for patients with cardiac implantable electronic devices has significantly improved physical activity. This study is designed as a prospective, single center, double-blind, randomized controlled trial. Divided into an experimental group and a control group at a ratio of 1:1. The experimental group with cardiac implantable electronic devices will receive cardiac rehabilitation health education video intervention, and the control group will receive only health education. We aim to recruit 45 participants per group with a total of 90 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-100 years old
* Patients with cardiovascular implantable electronic devices(CIEDs)
* CIEDs were implanted for more than 30 days without complications

Exclusion Criteria:

* cannot sign informed consent
* cannot return for follow-up visits current or scheduled enrollment in other conflicting studies
* concomitant disease (e.g., terminal cancer) or other medical condition likely to result in death within 6 months
* patients with bed-ridden status could not perform home-based tele-rehabilitation
* pregnancy

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Device measurement: physical activity | We collected data on the day of case enrollment and twelve weeks later.
  use CIEDs to measure, it shows as how many hours of physical activity a day.

SECONDARY OUTCOMES:
IPAQ, International Physical Activity Questionnaire | We collected data on the day of case enrollment and between 12 to 24 weeks later.
  The total physical activity score is calculated by summing the duration and frequency of vigorous, moderate, and walking activities. Higher scores indicate a higher physical activity.
SF-36, short-form 36 | We collected data on the day of case enrollment and between 12 to 24 weeks later.
  SF-36 is used to evaluate the "quality of life", range form 0-100. The survey results are interpreted in two main way: Domain Scores and Summary Scores. Higher scores represent better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Tsun Liao, PHD, Study Director — National Taiwan University Hospital Hsin-Chu Branch Hsinchu
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piepoli MF, Corra U, Adamopoulos S, Benzer W, Bjarnason-Wehrens B, Cupples M, Dendale P, Doherty P, Gaita D, Hofer S, McGee H, Mendes M, Niebauer J, Pogosova N, Garcia-Porrero E, Rauch B, Schmid JP, Giannuzzi P. Secondary prevention in the clinical management of patients with cardiovascular diseases. Core components, standards and outcome measures for referral and delivery: a policy statement from the cardiac rehabilitation section of the European Association for Cardiovascular Prevention & Rehabilitation. Endorsed by the Committee for Practice Guidelines of the European Society of Cardiology. Eur J Prev Cardiol. 2014 Jun;21(6):664-81. doi: 10.1177/2047487312449597. Epub 2012 Jun 20. PMID 22718797
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Pavy B, Iliou MC, Verges-Patois B, Brion R, Monpere C, Carre F, Aeberhard P, Argouach C, Borgne A, Consoli S, Corone S, Fischbach M, Fourcade L, Lecerf JM, Mounier-Vehier C, Paillard F, Pierre B, Swynghedauw B, Theodose Y, Thomas D, Claudot F, Cohen-Solal A, Douard H, Marcadet D; Exercise, Rehabilitation Sport Group (GERS); French Society of Cardiology. French Society of Cardiology guidelines for cardiac rehabilitation in adults. Arch Cardiovasc Dis. 2012 May;105(5):309-28. doi: 10.1016/j.acvd.2012.01.010. Epub 2012 Apr 16. No abstract available. PMID 22709472
- [Background] Mond HG, Proclemer A. The 11th world survey of cardiac pacing and implantable cardioverter-defibrillators: calendar year 2009--a World Society of Arrhythmia's project. Pacing Clin Electrophysiol. 2011 Aug;34(8):1013-27. doi: 10.1111/j.1540-8159.2011.03150.x. Epub 2011 Jun 27. PMID 21707667
- [Background] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Calabro MA, Kim Y, Franke WD, Stewart JM, Welk GJ. Objective and subjective measurement of energy expenditure in older adults: a doubly labeled water study. Eur J Clin Nutr. 2015 Jul;69(7):850-5. doi: 10.1038/ejcn.2014.241. Epub 2014 Nov 5. PMID 25351651